CLINICAL TRIAL: NCT02113384
Title: Prospective Observational Study of Exfoliated Peritoneal Tumor Cells in Locally Advanced Rectal Cancer
Brief Title: Locally Advanced Rectal Cancer - Exfoliated Peritoneal Tumor Cells
Acronym: LARC-EX
Status: Active, not recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Principal Investigator, Kjersti Flatmark, Professor, Oslo University Hospital
Other Study IDs: Larc-Ex_09/2012
Record Dates: First submitted 2014-04-08; First posted 2014-04-14 (Estimated); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer; Locally advanced rectal cancer; Peritoneal carcinomatosis; Exfoliated peritoneal cells; Peritoneal lavage
MeSH Terms: conditions — Rectal Neoplasms; Peritoneal Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Tumor tissue, peritoneal lavage samples, blood specimen.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational study: Patients with locally advanced rectum cancer undergoing surgical resection of the primary tumor at the Norwegian Radium Hospital.
  Interventions: Other: Observational study.

INTERVENTIONS:
Other: Observational study. — Biobanking of tissue (tumor biopsy, peritoneal lavage, blood specimen) from patients with locally advanced rectum cancer undergoing surgical resection of the primary tumor at the Norwegian Radium Hospital.
  Other Names: Observational study. Laboratory biomarker analysis.

SUMMARY:
During the course of tumor growth and possibly by manipulation during the surgical procedure, cells from rectal tumors may be shed into the peritoneal cavity. Such cells may give rise to local recurrence or contribute to the formation of metastatic disease, specifically in the form of peritoneal carcinomatosis. Detection of cancer cells in the peritoneal cavity at the time of surgery might therefore be of value for prediction of disease recurrence with subsequent prognostic implications for these patients. In this study the investigators aim to determine the presence of exfoliated tumor cells in peritoneal lavage samples from patients undergoing surgery for LARC.

DETAILED DESCRIPTION:
The investigators recently published a study investigating the incidence of exfoliated cancer cells in peritoneal lavage fluid after resection of locally advanced rectal cancer (LARC). DNA isolated from cells obtained by peritoneal lavage was analyzed by denaturing capillary electrophoresis with respect to mutations in hotspots of the K-RAS gene. This gene is mutated in 30% of rectal tumors. Exfoliated tumor cells (as assessed by the presence of mutated DNA) were found in lavage fluid from 19/237 of the patients, and the presence of tumor cells was associated with poor overall survival. Based on these encouraging results the investigators have designed a more comprehensive prospective study, using a novel, validated set of cancer specific DNA methylation - based biomarkers present in the vast majority of all colorectal tumors (sensitivity 94%, specificity 98%).Using these tumor cell associated biomarkers, the investigators aim to determine the presence of exfoliated tumor cells in peritoneal lavage samples from patients undergoing surgery for LARC. Lavage will be performed prior to and after manipulation of the tumor to provide data regarding both spontaneous and iatrogenic tumor cell exfoliation and their respective contribution to patient outcome. If detection of exfoliated tumor cells is predictive of tumor recurrence, this would support an active approach to postoperative chemotherapy, possibly in the form of intraperitoneal chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for surgical removal of a primary locally advanced rectal tumor at the Norwegian Radium Hospital.
* age > 18 years
* written informed consent

Exclusion criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for surgical removal of a primary locally advanced rectal tumor at the Radium Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 231 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years
  Time from surgery until death from any cause

SECONDARY OUTCOMES:
Disease-free survival | 5 years
  Time from surgery until disease recurrence or death
Disease-free survival | 3 years
  Time from surgery until disease recurrence or death
Overall survival | 3 years
  Time from surgery until death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Bjørn-Atle Bjørnbeth, MD PhD, Study Chair — Oslo University Hospital
Locations (1):
- The Norwegain Radium Hospital, Oslo, Ullern, Norway

IPD SHARING:
Plan to Share IPD: Undecided